CLINICAL TRIAL: NCT04202575
Title: Elimination of CO2-insufflation-induced Hypercarbia in Open Heart Surgery Using a Separate Reservoir for Suction of Blood From the Open Surgical Wound
Brief Title: Elimination of CO2-insufflation-induced Hypercarbia in Open Heart Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jan van der Linden, Professor, Karolinska University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018/1091-31
Record Dates: First submitted 2019-12-15; First posted 2019-12-17 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Adult Patients Undergoing Open Heart Replacement of the Aortic Valve for Aortic Stenosis or Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional setup (No Intervention): Blood and gas from the coronary and cardiotomy suction devices is continuously evacuated via the additional reservoir to the standard reservoir.
- Intervention setup (Experimental): The connecting tube between the additional and standard venous reservoir is clamped. Thus, blood and gas from the coronary and cardiotomy suction devices are collected in the additional venous reservoir. During the intervention setup, the blood in the additional venous reservoir is only evacuated to the standard reservoir if the volume exceeded 800ml, and always with a remaining volume of 100 mL blood to keep the CO2-gas trapped in the additional venous reservoir.
  Interventions: Procedure: Tube clamping

INTERVENTIONS:
Procedure: Tube clamping — Clamping of the tube between the additional and standard venous reservoir
  Arms: Intervention setup

SUMMARY:
The study aim was to evaluate if an additional separate venous reservoir eliminates CO2-insufflation induced hypercapnia and keeps sweep gas flow of the oxygenator constant during open heart surgery.

DETAILED DESCRIPTION:
Background: CO2-gas insufflation is used for continuous de-airing during open heart surgery. The study aim was to evaluate if an additional separate venous reservoir eliminates CO2-insufflation induced hypercapnea and keeps sweep gas flow of the oxygenator constant.

Methods: A separate small reservoir are used during CPB in addition to a standard large venous reservoir. The small reservoir receive drained wound blood and CO2-gas continuously via a suction drain (1 L/min) and handheld suction devices from the open surgical wound. CO2-gas is insufflated via a gas-diffuser in the open surgical wound at 10 L/min. During cross-clamping, gas and blood are either continuously drained to the standard large venous reservoir or not, every 5 minutes after steady state of PaCO2 is observed, after adjustment of sweep gas flow as necessary. Mean values for each setup (2-4 times) for each patient will be analyzed with Wilcoxon rank-sum test.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing open heart replacement of the aortic valve
* Use of perioperative cardiopulmonary bypass

Exclusion Criteria:

* Denied participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Difference in PaCO2 (kPa) | At 5 minutes steady state

SECONDARY OUTCOMES:
Oxygenator sweep gas flow rate (L/min) | At 5 minutes steady state

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
If other researchers would show interest in the data, we may considered providing data on a group level. However, individual data cannot be made available due to the rules in the GDPR.

REFERENCES:
- [Derived] Nyman J, Holm M, Fux T, Sesartic V, Fredby M, Svenarud P, van der Linden J. Elimination of CO2 insufflation-induced hypercapnia in open heart surgery using an additional venous reservoir. Interact Cardiovasc Thorac Surg. 2021 Aug 18;33(3):483-488. doi: 10.1093/icvts/ivab082. PMID 34363470